CLINICAL TRIAL: NCT03452566
Title: Phase 1/2 Clinical Trial for the Evaluation of Ingenol Mebutate for Actinic Cheilitis
Brief Title: Evaluation of Ingenol Mebutate for Actinic Cheilitis Treatment
Acronym: EIMAC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Ingenol mebutato discontinued in Brazil.
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 82279418.6.0000.5274
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Actinic Cheilitis
Keywords: actinic cheilitis; ingenol mebutate; treatment; phase 1/2 clinical trial
MeSH Terms: conditions — Actinic cheilitis | interventions — 3-ingenyl angelate

STUDY DESIGN:
Intervention Model Description: To determine the toxicity profile and the maximum tolerated dose (MTD) of ingenol mebutate for treatment of actinic cheilitis and to determine the therapeutic response with a dose below the maximum tolerated dose (MTD). The MTD will be tested in the phase 2 stage of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ingenol mebutate gel (Experimental): Phase 1/2, always 3 consecutive days, with 24 hours interval, dosage from 5 mg/cm2 to 18 mg/cm2 in a 3+3 design.
  Interventions: Drug: Ingenol mebutate gel

INTERVENTIONS:
Drug: Ingenol mebutate gel — 3+3 phase 1 design as described above. After the maximum tolerated dose is defined, the phase 2 segment of the study will take place. Simon's Phase 2 study design tool was used, reinforced by Jung's admissible study designs for phase 2 clinical trials. Considering the margin of error of 0.05 and study power of 80%, and estimating the probability of placebo partial response of 15% and partial response to ingenol mebutate in 45%, the optimized number of patients to be recruited is 19. Six patients will be seen in the first stage of this segment of the study, and if only one patient or none has a partial response, the study will be promptly discontinued. Otherwise, the second and final stage of segment of the study will include an additional thirteen patients who will be treated.
  Other Names: Picato

SUMMARY:
Actinic cheilitis is a major potentially carcinogenic disorder of the lower lip and several reports of clinical cases with excellent results for the treatment of this lesion that can differentiate to squamous cell carcinoma of the lip. However, clinical trials are lacking to define the optimal dosage of the drug for a therapeutic modality and to define its true efficacy in controlled studies of this pre-malignant labial lesion.

DETAILED DESCRIPTION:
Squamous cell carcinoma is the most common malignant neoplasm in the head and neck region, and when present in the lower lip, it is usually associated with prolonged exposure to UV radiation of lip vermilion surface especially in white patients (patients with genodermatosis such as xeroderma pigmentosum have extreme sensitivity to UV radiation, characterized by an even higher risk and patients presenting radiodermatites that can evolve to squamous cell carcinoma). Ingenol mebutate is a natural medicine derived from the sap of the pepense euphoria and much used for its medicinal properties.

The objective of this study was to determine the toxicity profile and the maximum tolerated dose (MTD) of ingenol mebutate for treatment of actinic cheilitis in patients of the Oncology Dermatology Session of the National Cancer Institute of Brazil (INCA) through a phase 1 clinical trial of type 3 + 3 and to determine the therapeutic response with a dose below the maximum tolerated dose (MTD) of metamato of ingenuity, for the treatment of aortic cheilitis in patients of the Oncology Dermatology Session of the National Cancer Institute (INCA) through a prospective clinical trial and phase randomized trial (phase 2).

Actinic cheilitis is a major potentially carcinogenic disorder of the lower lip and several reports of clinical cases with excellent results for the treatment of this lesion that can differentiate to squamous cell carcinoma of the lip. However, clinical trials are lacking to define the optimal dosage of the drug for a therapeutic modality and to define its true efficacy in controlled studies of this pre-malignant labial lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of actinic cheilitis .
* Histopathological report compatible with the clinical diagnosis.
* Sign the informed consent to be a part of the study.
* Comply with the attendance at the clinical settings during the days the patient will be medicated (D1, D2 and D3), D5, D8, two months, six months and one year after treatment.

Exclusion Criteria:

* Patients younger than 18 years of age.
* Patients without confirmed diagnosis of actinic cheilitis.
* Patients previously treated with ingenol mebutate for actinic cheilitis, including those in the present study, previously excluded at some point during phases 1 or 2.
* Presence of recurrent lesions, prior or during treatment.
* Immunosuppression.
* Use of topical corticosteroids.
* Presence of markedly hyperkeratotic or ulcerated lesions in the clinical evaluation
* Patients presenting with atypical histology (moderate to severe epithelial dysplasia) at the lips.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Female
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Actinic cheilitis response to treatment | Twelve months
  A 45% partial response to ingenol mebutate

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen Goldemberg, PhD, Principal Investigator — Researcher